CLINICAL TRIAL: NCT03259659
Title: Autonomic and Cytokines Profiles of Patients With Ulcerative Proctitis
Status: Terminated | Type: Observational
Why Stopped: Principal Investigator was leaving the institution.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00095405
Record Dates: First submitted 2017-08-21; First posted 2017-08-24 (Actual); Last update posted 2020-07-31 (Actual); Status verified 2019-09

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Microbiota

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — blood sample for inflammatory cytokines, fecal sample for microbiota
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- irritable bowel disease patient: Patients with ulcerative proctitis and proctosigmoiditis who meet the inclusion criteria, they will have ECG recording, inflammatory cytokines, microbiota, ulcerative colitis disease activity index.
  Interventions: Other: ECG recording, inflammatory cytokines, microbiota, ulcerative colitis disease activity index
- healthy control: Healthy participates who meet the inclusion criteria, they will have ECG recording, inflammatory cytokines, microbiota, ulcerative colitis disease activity index.
  Interventions: Other: ECG recording, inflammatory cytokines, microbiota, ulcerative colitis disease activity index

INTERVENTIONS:
Other: ECG recording, inflammatory cytokines, microbiota, ulcerative colitis disease activity index — In this study, an electrocardiogram signal will be recorded for 30 min in the fasting state, and blood samples for inflammatory cytokines analysis (7 ml) will be taken at the end of the ECG recording; fecal samples will be taken on the experimental day before the study. In addition, ulcerative colitis disease activity index will be assessed using the Mayo scoring system.

SUMMARY:
1. To prove that patients with ulcerative proctitis and proctosigmoiditis have impaired autonomic functions, i.e. increased sympathetic activity and/or reduced vagal tone.
2. To demonstrate inflammatory cytokine imbalance, i.e., increased pro-inflammatory cytokines. Presence of these abnormalities would make patients with ulcerative proctitis and proctosigmoiditis good candidates for future sacral nerve stimulation therapy.

ELIGIBILITY:
Inclusion Criteria:

* No any systemic diseases;
* no proctitis or proctosigmoiditis;
* no history of gastrointestinal surgery;
* no symptoms of diarrhea or fecal urgency during the past 2 weeks;
* not taking any medications except contraceptives during the past 2 weeks;
* age 18-65.

Exclusion Criteria:

* None.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: irritable bowel disease patients and healthy controls.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2020-02-29 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
symptoms characteristics in ulcerative colitis patients | 1 day
  ulcerative colitis disease activity index will be assessed using the Mayo scoring system, which includes stool frequency, rectal bleeding, mucosal appearance at endoscopy and physician rating of disease activity. The patient will get a score from 0 to 20, with higher score indicating more severe disease.

SECONDARY OUTCOMES:
autonomic profile characteristics in ulcerative colitis patients and healthy controls | 1 day
  heart rate variability indicating sympathetic and parasympathetic activity
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Granulocyte-colony stimulating factor (G-CSF)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Eotaxin
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Granulocyte-macrophage colony-stimulating factor (GM-CSF)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -1α
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Leptin
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Macrophage Inflammatory Proteins (MIP) -1α
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -4
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -1β
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -2
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -6
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Epidermal growth factor (EGF)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -13
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -10
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -12p70
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Interferon gamma (IFNγ)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -5
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -17A
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, interleukin (IL) -18
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Monocyte Chemoattractant Protein-1 (MCP-1)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Interferon - induced protein 10 (IP-10),
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, growth regulated oncogene (GRO)/Keratinocyte chemoattractant KC/cytokine-induced neutrophil chemoattractant (CINC)-1
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Vascular endothelial growth factor (VEGF)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Fractalkine
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Lipopolysaccharide-induced CXC chemokine (LIX)
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Macrophage Inflammatory Proteins (MIP) -2
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, Tumor necrosis factor (TNF) α
inflammatory cytokine profile in ulcerative colitis patients and healthy controls | 1 day
  blood sample, RANTES (Regulated on Activation, Normal T Cell Expressed and Secreted)
microbiota profile in ulcerative colitis patients and healthy controls | 1 day
  fecal sample microbiota analysis

CONTACTS AND LOCATIONS:
Overall Officials: Jiande Chen, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided